CLINICAL TRIAL: NCT06935461
Title: Families Moving Forward Bridges: An Early Intervention Enhancement for Infants and Toddlers With Prenatal Alcohol Exposure With or At-risk for Fetal Alcohol Spectrum Disorders
Brief Title: Families Moving Forward Bridges: An Early Intervention for Infants and Toddlers With PAE With or At-risk for FASD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Tracy Jirikowic, Professor, School of Medicine: Rehabilitation Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00020599; 1R61AA031695-01 (NIH)
Record Dates: First submitted 2025-03-14; First posted 2025-04-20 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Prenatal Alcohol Exposure; Fetal Alcohol Spectrum Disorders
Keywords: early childhood intervention; prenatal alcohol exposure; fetal alcohol spectrum disorder; infants and toddlers; FASD informed intervention
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FMF Bridges Early Intervention Program (Other): Following enrollment, a baseline assessment session will be completed (see caregiver and child assessments document uploaded). Following the assessment, the caregiver will receive intervention services from a trained FMF Bridges Specialists from Wonderland Child and Family Services within 1 month of completing the baseline assessment. The trained EI providers will deliver the FMF Bridges intervention, comprised of 10, 60-minute manualized intervention sessions (see FMF Bridges Intervention Protocol and Materials document). Sessions are expected to be delivered weekly or bi-weekly in the home (the standard of care for EI services), over a 3-to-5-month time period, with those electing to complete weekly sessions taking approximately 3 months or up to 5 for those who choose biweekly sessions. Outcome measures will be immediately post-intervention, as close as possible to the last session, and within 1 month of completing the intervention. Outcome measures at baseline and post interventio
  Interventions: Behavioral: Families Moving Forward Bridges

INTERVENTIONS:
Behavioral: Families Moving Forward Bridges — Ten, 60-minute manualized FMF Bridges intervention sessions over 3-5 months (approximately every other week)

SUMMARY:
This is an unblinded, feasibility study of an adapted positive parenting intervention to be carried out in a small sample (n=12 dyads) of young children with FASD and their primary caregiver in King County, WA.

DETAILED DESCRIPTION:
This is an initial feasibility study to examine Families Moving Forward Bridges (FMF Bridges), an FASD-informed early intervention designed to meet the specific needs of young children 6-36 months with prenatal alcohol exposure (PAE) or FASD and their caregivers. FMF Bridges was developed by this research team and is adapted from a scientifically-validated positive parenting intervention (Families Moving Forward) shown to be efficacious with preschool and school-aged children affected by PAE or FASD. FMF Bridges merges key components of FASD-informed care with family-centered and relationship-based early intervention practices and is designed to be delivered in community-based early intervention programs. The FMF Bridges early intervention needs to be tested with children and families in the community-based early intervention settings for which it was designed. The study team plans to evaluate the feasibility of FMF Bridges in a small community trial. the team will partner with an early intervention program that has a high population of children with prenatal alcohol exposure. EI providers will be trained as FMF Bridges Specialists and deliver the intervention to a total of 12 dyads (young child and their primary caregiver). Dyads will receive ten 60-minute manualized FMF Bridges intervention sessions over 3-5 months (approximately every other week) from community EI providers trained as FMF Bridges Specialists.

Primary Aim 1: Examine the feasibility of implementing the FMF Bridges early intervention in a community early intervention setting.

The study will focus on answering the questions: 1) Is it practical to implement the FMF Bridge intervention in a community EI setting? 2) Can the intervention be implemented with fidelity? 3) Is the intervention acceptable to providers and caregivers? and 4) What refinements might be needed to improve the feasibility of implementation?

ELIGIBILITY:
Inclusion Criteria:

* Child inclusion criteria: Infants and toddlers 6-36 months of age, any gender, any race/ethnicity, who:

  1. have confirmed PAE as ascertained by the standard child development center intake procedures;
  2. and 2) qualify for IDEA Part C EI services based on presence of a developmental delay (>25% in one or more areas of development) or therapist/provider informed clinical opinion.

Caregiver inclusion criteria:

1. biological, foster, adoptive, or other legal guardian;
2. age 18 or older;
3. any gender.

Exclusion Criteria:

* Child exclusion criteria:

  1. child has lived with current caregiver for less than 30% of chronological age or there is a planned change in caregiver placement or move out of King County within 3 months of intake;
  2. child has a medical or congenital/genetic condition that would severely limit participation in assessments, such as a significant visual or hearing impairment, degenerative muscle condition, or uncontrolled seizures;
  3. multiple birth;
  4. child currently receives inpatient medical care (e.g., NICU) or has a medical condition requiring a planned inpatient hospitalization or surgical intervention (e.g., heart condition);
  5. child diagnosis of a known genetic or non-FASD neurodevelopmental condition (e.g., Down syndrome, autism spectrum disorder).

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Devereux Early Childhood Assessment-Infant/Toddler (DECA-IT) | From enrollment to the end of intervention 3-5 months
  Standardized parent rating scale assessing child initiative, attachment, and self-regulation. Internal consistency (α=.90-.94); test-retest reliability (r= .91-.99).
Parenting Interactions with Children - Checklist of Observations Linked to Outcomes (PICCOLO) 86 | From enrollment to the end of intervention 3-5 months
  An observational measure of caregiver behavior including affection, responsiveness, encouragement, and teaching through caregiver-child interactions. Internal consistency (α=.75-.80); interrater reliability (r= .74-.80); construct validity (r= .62).
Family Outcomes Survey - Revised (FOS-R) | From enrollment to the end of intervention 3-5 months
  Designed to measure family outcomes and helpfulness of early intervention. Parent survey to rate the extent to which they have achieved family outcomes including knowing their rights and advocate effectively for their child, understand their child's strengths and needs, help their child develop and learn, have support systems, and access desired community services, programs, and activities.
Healthy Families Parenting Inventory (HFPI) | From enrollment to the end of intervention 3-5 months
  Designed to measure outcomes in home visitation programs. A survey of multiple dimensions of parenting: parent social support, problem solving, depression, personal care, mobilizing resources, role satisfaction, parent-child interactions, the home environment and parenting efficacy. Good internal consistency; evidence for convergent validity.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Jirikowic, PhD, Principal Investigator — University of Washington
Locations (1):
- Wonderland Child Development Center, Shoreline, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the statistical analysis plan. We will not share informed consent or study protocol because this is a feasibility study with a small sample.
Supporting Information: SAP, CSR
Time Frame: Data will become available after analysis is complete. Following the conditions and timeline in the NIMH data archive.
Access Criteria: Individual level data deidentified will be shared in the NIMH Data Archive.